CLINICAL TRIAL: NCT03986411
Title: Physiotherapy Management of Urinary Incontinence in Athletic Women- A Feasibility Study
Brief Title: Physiotherapy to Treat Urinary Incontinence in Athletes
Acronym: POsITIve
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: A2RMUR
Record Dates: First submitted 2019-06-10; First posted 2019-06-14 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2020-11

CONDITIONS: Urinary Incontinence
Keywords: urinary incontinence; pelvic floor; athlete
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: Mixed methods feasibility study. Three phases: Phase 1: Interviews Health car professionals, Phase 2: Intervention, Phase 3: Interviews of Participants
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Feasibility study of physiotherapy for UI in athletic women (Other): A mixed methods study with 3 distinct but related phases to explore the feasibility of conducting an RCT of physiotherapy as management of urinary incontinence in athletic women
  Interventions: Other: Phase 1: Qualitative interviews: Health care professionals; Other: Phase 2: Physiotherapy for urinary incontinence; Other: Phase 3: Qualitative Interviews: Participants

INTERVENTIONS:
Other: Phase 1: Qualitative interviews: Health care professionals — Semi-structured interviews of health care professionals to explore current management of urinary incontinence in the community
Other: Phase 2: Physiotherapy for urinary incontinence — Tailored physiotherapy assessment and management for athletic women who self-report urinary incontinence
Other: Phase 3: Qualitative Interviews: Participants — Semi-structured interviews of a purposeful selection of the participants from Phase 2 to explore reaction to the recruitment process and the intervention

SUMMARY:
Nearly half of all adult women suffer with Urinary incontinence (UI), this is more common in athletes.

UI is considered to be due to weak pelvic floor muscles. Standard advice encourages strength and endurance training; however, assessment of pelvic floor muscles can sometimes reveal overactive or tight tissues.

Evidence suggests athletes have stronger pelvic floors than non-athletes. If the pelvic floor is overactive, general advice regarding pelvic floor strengthening will not improve UI, and may make it worse.

This study will explore the feasibility of conducting a larger trial to identify cost effectiveness and benefits of treating athletes with physiotherapy and how this might differ from current practice.

15 -20 athletic women will complete questionnaires regarding their UI and its effects on them. They will receive physiotherapy; the assessment will include a history and internal examination of their pelvic floor. This will inform a tailored rehabilitation program.

Interviews will be conducted with some of these women to explore their response to the intervention. Interviews with health professionals will establish current practice for this patient group.

The results will tell us how likely it is for athletes to volunteer and take part in a future study and which outcomes are useful.

DETAILED DESCRIPTION:
Aims: The investigator's overall purpose is to conduct an RCT to determine whether one to one physiotherapy can improve the symptoms of urinary incontinence (UI) in a group of athletic women. This feasibility study will enable us to ascertain the viability of conducting a definitive appropriately powered trial.

Research protocol: The research design is a mixed methods study with three distinct but related phases.

Phase 1: 6-8 local health care professionals (GPs, nurses and physiotherapists) will be recruited for interview to explore current management practices of urinary incontinence (UI) in primary care.

Phase 2: 15-20 sporting or athletic women who self- report symptoms of UI will be recruited from the local sporting community. Each will undergo individual subjective and objective assessments in order to establish history, symptoms and pelvic floor muscle function. The intervention will be then be tailored from these assessments and agreed between each individual and the specialist physiotherapist. It will include guided exercise within the clinic and a regular home exercise plan, in keeping with typical pelvic health regimes for pelvic floor muscle (PFM) dysfunction.

Phase 3: 6-8 participants from phase 2 will be invited to take part in a qualitative interview in order to gain more in-depth understanding of UI. Purposeful selection will account for age, sporting activity and severity of symptoms. The interviews will be to explore the effects of UI on their quality of life, their participation in sport and exercise and the acceptability of the intervention.

Measurable end points: 6 months from recruitment of the last participant in phase 2 will be considered to be the end point of the study.

ELIGIBILITY:
Inclusion Criteria:

* Phase 1: Qualified local Health Care Professional eg G.P., nurse or chartered physiotherapist working within Nottinghamshire or Derbyshire
* Phases 2 and 3:Adult female Currently exercising for a minimum 3 times a week and for over 150 minutes per week Self-reported experience of symptoms of UI defined as; leaking of urine associated with increased abdominal pressure e.g. impact, leaking of urine associated with urinary urge, increased urinary urge and/or increased urinary frequency

Exclusion Criteria:

* Phase 1: Unwilling or unable to provide written informed consent Not within Nottinghamshire or Derbyshire area
* Phases 2 and 3: Under 18 Sports participation less than 1 year Pregnancy Less than one year after childbirth Ongoing physiotherapy or continence advice treatment elsewhere or within the last year De novo oestrogen or anticholinergic treatment Existing neurological conditions that may contribute to UI eg multiple sclerosis, stroke, spinal injury etc Unwilling or unable to provide written informed consent Unable to read or speak English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-08-27 (Actual); Primary Completion 2020-12-03 (Actual); Study Completion 2020-12-03 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | Up to 8 Months
  Ease of recruiting participants directly from gyms and sports clubs
Attrition rate | 6 months after the participant's first assessment
  The number of participants who consent to participate that remain in the study
Acceptability of the intervention: % that give positive feedback from the interviews | Up to 9 months
  Measured as the % that give positive feedback from the interviews in Phase 3
Acceptability of the secondary outcome measures used in Phase 2: % positive feedback for each outcome measure from the interviews | Up to 9 months
  Measured as the % positive feedback for each outcome measure from the interviews in Phase 3
Timescale required for intervention | Six months for each participant from the first assessment
  The time required for a successful intervention. This will be measured by the change in the secondary outcome measures between the three month assessment and the six months assessment

SECONDARY OUTCOMES:
Urinary Distress Inventory (UDI) 6 | Six months from the first assessment for each participant
  A short questionnaire to evaluate 'bother' of urinary symptoms (6 questions) mean score x 33.3 to give a final score out of 100. Where 100 indicates the most severe urinary distress
International Consultation on Incontinence Modular Questionnaire Female Lower Urinary Tract Symptoms Long Form Module (ICIQ-FLUTS-LF) | Six months from the first assessment for each participant
  A long quality of life and descriptive questionnaire to establish type and severity of urinary symptoms and the impact of these on quality of life (Two scores: urinary symptoms max score 69 where this is indicates the most severe; quality of life score, where the maximum score is 150, where urinary symptoms are having the maximum negative impact on quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Gillian Campbell, BVMS BSc PhD, Principal Investigator — University of Nottingham
Locations (1):
- University of Nottingham, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data may be made available to other researchers at the end of the study
Supporting Information: Study Protocol, ICF
Time Frame: 31/01/2021 for up to 5 years
Access Criteria: By direct contact to the study PI

REFERENCES:
- [Derived] Campbell KG, Nouri F, E Batt M, Drummond A. Management of urinary incontinence in athletic women: the POsITIve feasibility study. Physiotherapy. 2022 Mar;114:30-37. doi: 10.1016/j.physio.2021.12.001. Epub 2021 Dec 18. PMID 35101711
- [Derived] Campbell KG, Batt ME, Drummond A. A feasibility study of the physiotherapy management of urinary incontinence in athletic women: trial protocol for the POsITIve study. Pilot Feasibility Stud. 2020 Jul 16;6:103. doi: 10.1186/s40814-020-00638-6. eCollection 2020. PMID 32695435

DOCUMENTS (2):
  • Study Protocol (2019-03-28): https://cdn.clinicaltrials.gov/large-docs/11/NCT03986411/Prot_000.pdf
  • Informed Consent Form (2019-03-28): https://cdn.clinicaltrials.gov/large-docs/11/NCT03986411/ICF_001.pdf